CLINICAL TRIAL: NCT03801902
Title: Phase I Trial of Radiotherapy Combined With Durvalumab Alone Plus Either Monalizumab or Oleclumab in PD-L1 High Locally Advanced Non-Small Cell Lung Cancer (NSCLC) (ARCHON-1)
Brief Title: Testing the Safety of Adding Either Monalizumab (IPH2201) or Oleclumab (MEDI9447) to Durvalumab (MEDI4736) Plus Standard Radiation Therapy for Locally Advanced Non-small Cell Lung Cancer (NSCLC), ARCHON-1 Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00176; NCI-2019-00176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU004 (Other: NRG Oncology); NRG-LU004 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Locally Recurrent Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; durvalumab; Immunoglobulin G; Disulfides; Contrast Media; monalizumab; NK Cell Lectin-Like Receptor Subfamily C; Antibodies, Monoclonal, Humanized; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (CLOSED) (Durvalumab and ACRT) (Experimental): Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ACRT 1 fraction per day, 5 days per week for 15 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.
  Interventions: Radiation: Accelerated Hypofractionated Radiation Therapy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast
- Arm II (CLOSED) (Durvalumab and standard RT) (Experimental): Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast; Radiation: Radiation Therapy
- Arm III (durvalumab, monalizumab, standard RT) (Experimental): Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes and monalizumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast; Biological: Monalizumab; Radiation: Radiation Therapy
- Arm IV (durvalumab, oleclumab, standard RT) (Experimental): Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Patients also receive oleclumab IV over 60 minutes on days 1 and 15 of cycles 1-2, then on day 1 of cycles thereafter. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast; Biological: Oleclumab; Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Accelerated Hypofractionated Radiation Therapy — 160 Gy given as one 4 Gy fraction per day, 5 days per week for 15 fractions.
  Other Names: AHF-RT; AHRT
  Arms: Arm I (CLOSED) (Durvalumab and ACRT)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo brain CT and chest CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Administered intravenously (IV) as a 1500 mg fixed dose over 60 minutes for 13 cycles (1 cycle = 4 weeks), until disease progression or toxicity or death, whichever comes first.
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast — Undergo brain MRI
  Other Names: Brain Magnetic Resonance Imaging with and without Contrast; Brain MRI; Brain MRI with and without Contrast; Head MRI with and without Contrast
Biological: Monalizumab — Administered IV as a 1500 mg fixed dose over 60 minutes (+/- 10 minutes)
  Other Names: Immunoglobulin G4-kappa, Anti-(Homo sapiens KLRC1 (Killer Cell Lectin-like Receptor Subfamily C Member 1, NKG2-a, NKG2a, CD159A, CD94)), Humanized Monoclonal Antibody; IPH-2201; IPH2201; NN-8765; NN8765; NN8765-3658
  Arms: Arm III (durvalumab, monalizumab, standard RT)
Biological: Oleclumab — Administered IV 3000 mg over 60 minutes (+/- 10 minutes)
  Other Names: Anti-CD73 Monoclonal Antibody MEDI9447; MEDI9447
  Arms: Arm IV (durvalumab, oleclumab, standard RT)
Radiation: Radiation Therapy — 60 gy given as one 2 Gy fraction per day, 5 days per week for 30 fractions
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm II (CLOSED) (Durvalumab and standard RT); Arm III (durvalumab, monalizumab, standard RT); Arm IV (durvalumab, oleclumab, standard RT)

SUMMARY:
This phase I trial studies the safety of adding durvalumab to accelerated hypofractionated radiation therapy (ACRT) or conventionally fractionated radiation therapy, as well as the safety of adding either monalizumab or oleclumab to durvalumab plus conventionally fractionated radiation therapy in treating patients with non-small cell lung cancer that has spread to nearby tissue or lymph nodes (locally advanced). Accelerated hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Immunotherapy with monoclonal antibodies, such as durvalumab and monalizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Oleclumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD73, which is found on some types of tumor cells. Oleclumab may block CD73 and help the immune system kill tumor cells. It is not yet known whether adding durvalumab to ACRT or adding monalizumab or oleclumab to durvalumab plus conventionally fractionated radiation therapy will work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if the addition of durvalumab to two schedules of radiation therapies (60 Gy in 30 fractions or 60 Gy in 15 fractions) is safe.

II. To evaluate if the addition of either monalizumab or oleclumab to radiation therapy (RT) (60 Gy in 30 fractions) + durvalumab is safe.

SECONDARY OBJECTIVES:

I. To examine if the addition of durvalumab to radiation therapy as well as the addition of either monalizumab or oleclumab is feasible.

II. To assess toxicities associated with the addition of durvalumab to radiation therapy as well as the addition of either monalizumab or oleclumab.

III. To obtain preliminary estimates of progression-free survival (PFS), using Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, in patients who received durvalumab added to radiation, and either monalizumab or oleclumab added to RT (60 Gy in 30 fractions) + durvalumab.

EXPLORATORY OBJECTIVES:

I. To assess the impact the addition of durvalumab to RT and either monalizumab or oleclumab to RT (60 Gy in 30 fractions) + durvalumab have on progression-free survival, using Immune-Related Response Criteria (irRC) guidelines.

II. To assess the changes in circulating tumor cells (CTCs) and various immune parameters during treatment with durvalumab and radiotherapy and changes after completion of treatment.

OUTLINE: Patients are randomized to Arm I or Arm II (CLOSED TO ACCRUAL).

ARM I (CLOSED): Starting 2 weeks prior to radiation therapy, patients receive durvalumab intravenously (IV) over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo accelerated hypofractionated radiation therapy (ACRT) 1 fraction per day, 5 days per week for 15 fractions. Patients also undergo brain magnetic resonance imaging (MRI) or computed tomography (CT) scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.

ARM II (CLOSED): Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.

Patients are assigned to Arm III or Arm IV.

ARM III: Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes and monalizumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.

ARM IV: Starting 2 weeks prior to radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Patients also receive oleclumab IV over 60 minutes on days 1 and 15 of cycles 1-2, then on day 1 of cycles thereafter. Treatment repeats every 4 weeks for 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo conventionally fractionated radiation therapy 1 fraction per day, 5 days per week for 30 fractions. Patients also undergo brain MRI or CT scan during screening and as clinically indicated, chest CT scans on study and during follow up, and collection of blood samples during screening and on study.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic (cytological or histological) proof of diagnosis of stage II-III (American Joint Committee on Cancer [AJCC] 8th edition [ed.]) unresectable or inoperable, non-metastatic non-small cell lung cancer (NSCLC) within 60 days prior to registration, with no liver or renal end organ damage, as determined by normal laboratory values noted below. Locally recurrent, N1-N3 disease following surgery without prior radiation therapy is eligible. Patients with N1 to N3 and undetectable primary lung tumors (T0) are eligible
* Pathological diagnosis of PD-L1 high expressing tumors (>= 50%) within 60 days prior to registration (using Dako 22C3 immunohistochemistry [IHC] antibody or the Ventana SP263 antibody platforms) performed at a Clinical Laboratory Improvement Act (CLIA)-certified lab
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 30 days prior to registration;
  * Positron emission tomography (PET)/computed tomography (CT) scan for staging within 30 days prior to registration (note: if CT portion of PET/CT scan is not of diagnostic quality, then a separate CT scan with contrast is required);
  * Magnetic resonance imaging (MRI) scan of the brain with contrast; if medically contraindicated, then CT scan of the brain with contrast (unless medically contraindicated) is acceptable, within 30 days prior to registration;
  * Sufficient lung function with forced expiratory volume in 1 second (FEV1) >= 0.8 liter or >= 35% predicted and carbon monoxide diffusing capability (DLCO) >= 40% with or without bronchodilator within 30 days prior to registration;
  * Patients who meet the criterion above without oxygen (O2), but who need acute (started within 10 days prior to registration) supplemental oxygen due to tumor-caused obstruction/hypoxia are eligible, provided the amount of the O2 needed has been stable
* Age ≥ 18
* Minimum body weight >= 40 kg
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 (within 30 days prior to registration)
* Lymphocyte count >= 500 cells/mm^3 (within 30 days prior to registration)
* Platelet count >= 100,000 cells/mm^3 (within 30 days prior to registration)
* Hemoglobin >= 9.0 g/dL (within 30 days prior to registration) (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable)
* Creatinine clearance >= 40 mL/min by the Cockcroft-Gault (C-G) equation
* Total bilirubin =< 1.5 x upper limit of normal (ULN) with the following exception (within 30 days prior to registration):

  * Patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (within 30 days prior to registration)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients, obtained within 14 days prior to registration. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have a CD4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease
* Prior invasive malignancy (except those with a negligible risk of metastasis or death and with expected curative outcome [such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent] or undergoing active surveillance per standard-of-care management [e.g., chronic lymphocytic leukemia (CLL) Rai stage 0, prostate cancer with Gleason score =< 6, and prostate specific antigen (PSA) =< 10 mg/mL]) unless disease free for a minimum of 3 years
* Prior chemotherapy or systemic therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields so that cumulative composite dose combining previous plan and current plan to be within 80 Gy to the trachea, major blood vessels, esophagus, and heart, and 55 Gy to the spinal cord (if such patients are being considered, this will need to be centrally reviewed). Prior chest radiation without overlap is permissible
* Prior history of myocardial infarction, stroke, or transient ischemic attack in the past 3 months
* History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of treated autoimmune thyroid disease requiring thyroid replacement but not immunosuppressives, as well as type 1 diabetes, are permitted. Patients with vitiligo, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on chest PET/CT or CT scan
* Severe, active co-morbidity defined as follows:

  * Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease;
  * Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications;
  * Active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice);
  * Active hepatitis B (chronic or acute) or hepatitis C infection. Patients with past or resolved hepatitis B infection defined as having a negative hepatitis B surface antigen (HBsAg) test, a positive anti-HBc (antibody to hepatitis B core antigen), and a negative viral deoxyribonucleic acid (DNA) test (only obtained if HBsAg is found positive) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for 3 months after the last dose of treatment; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Women who are breastfeeding and unwilling to discontinue
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
* Major surgical procedure (as defined by the investigator) within 28 days prior to registration

  * Note:

    * Local surgery of isolated lesions for palliative intent is acceptable
    * Other major surgery before first dose of immunotherapy is not acceptable
* History of allogenic organ transplantation
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Current or prior use of immunosuppressive medication within 14 days before registration. (Note: immunosuppressive medication within 14 days before immunotherapy is not acceptable). The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to registration
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, Principal Investigator — NRG Oncology
Locations (56):
- United States (56):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT) | Arm III (Durvalumab, Monalizumab, Standard RT) | Arm IV (Durvalumab, Oleclumab, Standard RT)
Started | 14 | 12 | 0 | 0
Analyzable for Safety Events (Death or consent withdrawal within the safety monitoring period and before experiencing a safety event excludes a participant from this population.) | 12 | 12 | 0 | 0
Completed | 13 | 12 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Did not receive protocol treatment. | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Median (Full Range); unit: years] | 69 [53 to 78] | 72 [54 to 79] | 69 [53 to 79]
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 1 | 1 | 2
  60-69 years | 9 | 4 | 13
  ≥ 70 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 8 | 10 | 18
    1 | 5 | 2 | 7
Programmed death-ligand 1 (PD-L1) Value [Count of Participants; unit: Participants] — Programmed death-ligand 1 (PD-L1) is a protein that in humans is encoded by the CD274 gene. A PD-L1 test measures what percentage of cells in a tumor "express" PD-L1. Tumors that express high amounts of PD-L1 (50% or greater) may respond particularly well to checkpoint inhibitors.
  Participants
    50%-60% | 2 | 4 | 6
    70%-80% | 6 | 3 | 9
    >80% | 5 | 5 | 10
American Joint Committee on Cancer (AJCC) 8th ed. Stage [Count of Participants; unit: Participants] — Overall AJCC cancer stage combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively.
  Participants
    IIIA | 6 | 3 | 9
    IIIB | 4 | 7 | 11
    IIIC | 2 | 2 | 4
    N1-Undectable primary | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Safety Event
Description: Safety event is defined as one of the following:
  * Grade 4-5 non-hematologic protocol-defined serious adverse event (SAE) possibly, probably, or definitely related to protocol treatment occurring within 90 days from radiation therapy (RT) start for Arm 1 or within 8 weeks from RT start for Arm 2;
  * Any adverse event possibly, probably, or definitely related to protocol treatment that leads to missing at least 2 doses of durvalumab within 90 days from RT start for Arm 1 or within 8 weeks from RT start for Arm 2;
  * Permanent discontinuation of durvalumab due to an adverse event possibly, probably, or definitely related to protocol treatment within the first 30 days of starting durvalumab; or
  * SAEs possibly, probably, or definitely related to RT that cause either an interruption or early termination of RT.
  Adverse events are graded according to the Common Terminology Criteria for Adverse Events version 5.0, which assigns a grade according to severity from 1=mild to 5=death.
Time Frame: From start of study treatment to 90 (ACRT) or 56 (standard RT) days from the end of radiation treatment. (Approximately 104 or 70 days, respectively, from start of study treatment)
Population: Analyzable for safety events
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1
Statistical Analysis 1: Comparison: Arm I (CLOSED) (Durvalumab and ACRT) vs Arm II (CLOSED) (Durvalumab and Standard RT); Test type: Other; If 0-1 of initial 6 evaluable patients on an arm have a safety event, then the regimen will be deemed safe and that arm will continue to the second part of the study to enroll 6 additional evaluable patients. However, if 2 or more of the 6 patients develop a safety event, then that arm is considered not safe and will not continue to second part. The probability of the treatment being judged to be too toxic when the true toxicity rate is ≥ 40% is at least 77%. If the true toxicity rate is ≤ 18%, then the probability that the treatment will be deemed to be safe is at least 70%. If fewer than 4 of the total of 12 evaluable patients on an arm experience a safety event, then the treatment will be considered tolerable. With a cohort of 12 patients, the probability of the treatment being judged to be too toxic when the true toxicity rate is ≥ 40% at least 78%. If the true toxicity rate is ≤ 18%, the probability that the treatment will be deemed to be safe is 85%

2. Secondary Outcome: Percentage of Participants Who Received at Least 80% of Planned Durvalumab Dose During First 8 Weeks Following Initial Dose
Time Frame: From start of durvalumab to 8 weeks
Population: Eligible participants accrued to arm I or arm II.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
Number analyzed (Participants) | 13 | 12
percentage of participants | 84.6 [54.6 to 98.1] | 75.0 [42.8 to 94.5]

3. Secondary Outcome: Percentage of Participants Who Received at Least 80% of Planned Dose of Monalizumab or Oleclumab During the First 8 Weeks Following the Initial Dose (Feasibility)
Description: An observation of at least 80% of patients who received at least 80% of the planned dose is considered to be evidence that the given regimen is feasible in this setting.
Time Frame: From start of monalizumab or oleclumab to 8 weeks
Population: Eligible participants on arms III and IV. No participants accrued to these arms.
Arm/Group | Arm III (Durvalumab, Monalizumab, Standard RT) | Arm IV (Durvalumab, Oleclumab, Standard RT)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Distribution of Participants by Highest Grade Adverse Event
Description: Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 grades adverse event severity from 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From registration to last follow-up at time of initial analysis. Maximum follow-up was 23.2 months
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
Number analyzed (Participants) | 13 | 12
Participants
  Grade 1 | 2 | 0
  Grade 2 | 5 | 3
  Grade 3 | 4 | 8
  Grade 4 | 1 | 0
  Grade 5 | 1 | 1

5. Secondary Outcome: Percentage of Participants Experiencing a Grade 4 or Higher Non-hematologic Adverse Event
Description: as for outcome 4
Time Frame: From registration to last follow-up at time of initial analysis. Maximum follow-up was 23.2 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
Number analyzed (Participants) | 13 | 12
percentage of participants | 7.7 [0.2 to 36.0] | 8.3 [0.2 to 38.5]

6. Secondary Outcome: Progression-free Survival
Description: Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as an increase >= 20% of the sum of longest diameters of target lesions compared with nadir (minimum 5 mm) or progression of non-target lesions or new lesion. Progression-free survival time is defined as time from registration to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. Analysis was planned to occur two years after end of protocol treatment, which could last up to 12 months. No formal testing was planned due to a lack of statistical power.
Time Frame: From registration to two years after protocol treatment, which lasted up to 12 months. Maximum follow-up was 38.3 months.
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
Number analyzed (Participants) | 13 | 12
months | 20.4 [7.9 to NA] — There here were not enough events to estimate the upper confidence boundary. | 30.2 [8.2 to NA] — There here were not enough events to estimate the upper confidence boundary.

ADVERSE EVENTS:
Time Frame: From registration to two years after protocol treatment, which lasted up to 12 months. This time frame corresponds to the last outcome measure analyzed, progression-free survival.
Arm/Group | Arm I (CLOSED) (Durvalumab and ACRT) | Arm II (CLOSED) (Durvalumab and Standard RT)
All-Cause Mortality (participants affected / at risk) | 4/13 | 2/12
Serious Adverse Events (participants affected / at risk) | 6/13 | 5/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CLOSED) (Durvalumab and ACRT) (N=13) | Arm II (CLOSED) (Durvalumab and Standard RT) (N=12)
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Cardiac troponin T increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CLOSED) (Durvalumab and ACRT) (N=13) | Arm II (CLOSED) (Durvalumab and Standard RT) (N=12)
Anemia (Blood and lymphatic system disorders) | 4 | 6
Atrial fibrillation (Cardiac disorders) | 1 | 2
Palpitations (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 4
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 5 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 4
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 2
Fatigue (General disorders) | 12 | 9
General disorders and administration site conditions - Other (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 2
Pain (General disorders) | 1 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 1
Shingles (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 4
Alkaline phosphatase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 2 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0
INR increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 5 | 8
Platelet count decreased (Investigations) | 2 | 0
Thyroid stimulating hormone increased (Investigations) | 1 | 1
Weight loss (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 2
Stroke (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Psychiatric disorders - Other (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The study opened with 2 cohorts. Results were entered in 01-2022 and approved, after which the protocol was amended to add 2 cohorts such that the primary completion date (PCD) was changed to a future date, requiring entered results to be removed. The new cohorts opened accrual 01-2024. About a year later the decision was made to permanently close accrual. There was no accrual to the new cohorts, therefore PCD reverted to the prior date and the original outcome measure results were re-entered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2011-11-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT03801902/Prot_SAP_001.pdf
  • Informed Consent Form: PNRG-LU004_A13ConsentCohorts#1-4(Redacted) (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03801902/ICF_002.pdf
  • Informed Consent Form: PNRG-LU004_A13ConsentCohorts#5-8(Redacted) (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03801902/ICF_003.pdf